CLINICAL TRIAL: NCT01981902
Title: Non-Invasive Optical Spectroscopic Methods for Dehydration Identification in Marathon Trainees
Status: Withdrawn | Type: Observational
Why Stopped: Not a clinical trial study
Sponsor: University of California, Irvine (Other)
Collaborators: Beckman Laser Institute University of California Irvine (Other)
Responsible Party: Principal Investigator, Beckman Laser Institute and Medical Center, Matthew Brenner, M.D.,Department of Pulmonary and Critical Care Medicine, University of California, Irvine
Other Study IDs: 20129075
Record Dates: First submitted 2013-08-13; First posted 2013-11-13 (Estimated); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Dehydration
Keywords: Dehydration
MeSH Terms: conditions — Dehydration

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Dehydration: Non-Invasive Optical Spectroscopic monitoring method for dehydration
  Interventions: Device: Non-Invasive Optical Spectroscopic

INTERVENTIONS:
Device: Non-Invasive Optical Spectroscopic — Non-Invasive Optical Spectroscopic

SUMMARY:
Dehydration can result from exposure to harsh environments including hot and dry desert climates. Soldiers and non-military workers are frequently required to work in hot, dry conditions, and dehydration can be productivity limiting and life threatening if unrecognized.

DETAILED DESCRIPTION:
The research can use low power laser technology to take measurements of muscle tissue water content in volunteers before and after marathon training runs to detect dehydration. Two slightly different devices can be used to detect dehydration. 1). diffuse optical spectroscopy and 2). spatial frequency domain imaging-modulated imaging The researchers can determined by use other methods to assess the level of dehydration status in runners. These methods will include taking weight and temperature before and after run, skin-fold measurements pre and post run, and obtaining saliva samples from before and after run. The researchers can determine the study use non-invasive, laser light technology measure tissue water concentrations, as an indicator of dehydration.

ELIGIBILITY:
Inclusion Criteria:

* male female ages of 18 and 60
* training for a marathon

Exclusion Criteria:

1. Poorly controlled diabetes mellitus
2. Diabetes insipidus (excessive urination of water) as diagnosed by your physician
3. disorder of the intestine
4. Irritable bowel syndrome with excessive diarrhea, as diagnosed by a physician
5. Congestive heart failure and subsequent use of a diuretic "water pill" to remove excess water from the body
6. Have poor kidney function
7. Have been diagnosed with hyperthyroidism/hypothyroidism by your physician

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Study population are the volunteers who are training for a marathon individually or under the guidance of the Leukemia Society Team in Training, the American Heart Association, or similar groups. These organizations run programs that include providing group-training situations for individuals interested in preparing for a marathon while participating in fund raising efforts.
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2013-08; Primary Completion 2018-08 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Hydration | up to 4 weeks
  Marathon Trainees

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Brenner, MD, Principal Investigator — Beckman Laser Institute
Locations (1):
- Beckman Laser Institute University of California Irvine, Irvine, California, United States